CLINICAL TRIAL: NCT01332877
Title: The Effect of Breakfast Enriched With Protein and Carbohydrates on Weight Loss, Hunger, Satiety and Ghrelin in Overweight and Obese Adults
Brief Title: Breakfast Size and Weight Loss in Overweight/Obese Adults
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Prof. Daniel Jakubowicz, E. Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0029-11-WOMC
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; Ghrelin; Satiety; Hunger
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- enriched breakfast (Experimental): high carbohydrate, high protein breakfast providing 600 kcal, 50% carbohydrate, 20% protein, 30% fat
  Interventions: Behavioral: Enriched breakfast; Behavioral: Control breakfast

INTERVENTIONS:
Behavioral: Enriched breakfast — high carbohydrate, high protein breakfast supplying 600 kcal as 50k% carbohydrate, 20% protein, 30% fat
Behavioral: Control breakfast — Control breakfast providing 300 kcal, 13% carbohydrate, 40% protein, 48% fat

SUMMARY:
EFFECT OF HIGH CARBOHYDRATE AND HIGH PROTEIN BREAKFAST ON WEIGHT LOSS, GHRELIN, HUNGER AND CRAVING SCORES IN OBESE MEN AND WOMEN. D Jakubowicz, M Boaz, J Wainstein, O Froy

Background: Obesity underlying endocrine, metabolic and eating behaviour features promotes weight gain, increase of hunger, and carbohydrate (Carb) craving. Restrictive diets either in calories or Carb produce withdrawal effect, that further exacerbate Carb craving resulting in rapid return of obesity. Meal timing and composition has shown to play a pivotal role in appetite regulation through several hormonal systems such as ghrelin. The investigators hypothesized that to be successful; a weight loss strategy must change the hormonal environment to increase satiety while reducing hunger and craving.

Objectives: To assess weight loss, satiety, hunger, cravings and ghrelin response to two isocaloric diets. Additionally, these outcomes were measured in response to meal challenge.

Methods: In this randomized, treatment controlled clinical trial, 146 obese, sedentary adults with impaired glucose tolerance will be assigned to Low carb diet (LCHbd) or an isocaloric diet with a high carb, high protein breakfast (HCPbd),1400 kcal for women and 1600 kcal for men. LCHbd breakfast will provide 300 kcal with carb: protein: fat of 13:40:48. HCPbd breakfast will provide 600 kcal with 50:20:30. From baseline until week 16 participants will take part in a supervised weight loss diet, followed until week 32 by a maintenance period. Anthropometric measures, OGTT for glucose and insulin, VAS-measured hunger and satiety and Food Craving Inventory Analysis will be performed at baseline, week 16 and week 32.

ELIGIBILITY:
Inclusion Criteria:

* adult
* male and female
* obese
* sedentary
* glucose intolerant/insulin resistant

Exclusion Criteria:

* pregnant/lactating
* malignancy
* taking weight loss medications
* know eating disorder

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 32 weeks
  Change from baseline weight

SECONDARY OUTCOMES:
Hunger | 32 weeks
  VAS hunger scores
Satiety | 32 weeks
  VAS satiety scores
plasma ghrelin | 32 weeks
  change from baseline ghrelin

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Medical Center, Holon, Israel